CLINICAL TRIAL: NCT05464277
Title: Impact of Intermediate Normal Compared to High Normal Oxygen Levels on Outcomes of Patients Presenting in the Emergency Department With Severe Traumatic Brain Injury (INACHOS): a Pilot Randomized Controlled Trial
Brief Title: Intermediate Normal Versus High Normal Oxygen Levels in the Emergency Department for Severe Traumatic Brain Injury
Acronym: INACHOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient rate of recruitment
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Ilias Siempos, Academic Scholar, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 286/18-6-2020
Record Dates: First submitted 2022-07-10; First posted 2022-07-19 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Traumatic Brain Injury; Acute Respiratory Failure; Acute Respiratory Distress Syndrome; Acute Brain Injury
Keywords: emergency care; acute respiratory failure; trauma; oxygen; disability; acute care; critical care; mortality; brain injury; mechanical ventilation
MeSH Terms: conditions — Brain Injuries, Traumatic; Respiratory Distress Syndrome; Brain Injuries; Wounds and Injuries | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be randomly allocated using opaque sealed envelopes to either "intermediate normal oxygen" or "high normal oxygen" group. The asymptomatic maximal procedure, with an allocation ratio of 1:1 and a maximum tolerated imbalance of 2 will be used to randomize subjects.
Who Masked: Participant, Outcomes Assessor
Masking Description: To avoid selection bias, the allocation sequence will be blinded from researchers involved in patient enrolment. Although study subjects will be unaware of the assigned group, blinding of treating clinicians is not considered feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermediate normal oxygen (Active Comparator): For the "intermediate normal oxygen" group, an oxygen saturation by pulse oximetry (SpO2) of 95-97% will be recommended in the light of the Improving Oxygen Therapy in Acute-illness (IOTA) meta-analysis. The acceptable lower limit of PaO2 will be set to 80 mmHg according to a recent consensus of experts endorsed by the European Society of Intensive Care Medicine. The lower-limit and higher-limit monitor alarm for SpO2 will be set at 94% and 98%, respectively.
  In case that the emergency department of a study site uses ventilators, which allow for only two options of FiO2 titration (namely, "air mix" and "FiO2 of 1.0"), then the "intermediate normal oxygen" group should receive "air mix".
  Interventions: Other: Oxygen
- High normal oxygen (Active Comparator): For the "high normal oxygen" group, an oxygen saturation by pulse oximetry (SpO2) of 99-100% will be recommended. The lower-limit monitor alarm for SpO2 will be set at 98%. No upper alarm limit for SpO2 will be set.
  In case that the emergency department of a study site uses ventilators, which allow for only two options of FiO2 titration (namely, "air mix" and "FiO2 of 1.0"), then the "high normal oxygen" group should receive "FiO2 of 1.0".
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: Oxygen — Oxygen to achieve assigned SpO2 (or FiO2) targets will be administered to study subjects. The treating clinician can alter oxygenation targets at any time if deemed necessary. The oxygenation goal will be based on SpO2 rather than arterial oxygen saturation (SaO2) or arterial pressure oxygen (PaO2) from arterial blood gases. However, PaO2 can be used instead in situations where the treating clinician considers that peripheral perfusion is poor or SpO2 readings are unreliable. Assigned SpO2 targets will apply to the study subjects for a total duration of 6 hours from intubation or until death or until transfer to the operating theater (whatever comes first).

SUMMARY:
Despite almost universal usage of supplemental oxygen therapy in patients presenting in the emergency department with traumatic brain injury (TBI), optimal oxygen levels are unclear.

The investigators propose a pilot multi-center randomized controlled trial to test the hypothesis that maintaining intermediate normal as opposed to high normal oxygen levels in patients presenting in the emergency department with TBI is feasible, and to obtain preliminary data on the efficacy of the two approaches to oxygen therapy. The aim is that the investigators produce pilot data, which could inform the design of potential subsequent larger clinical trials.

DETAILED DESCRIPTION:
Despite the worldwide burden of traumatic brain injury (TBI), medical research on the field as opposed to other health problems is underrepresented. Consequently, there are few data to support commonly used interventions for the management of TBI, especially in the setting of the emergency department. For example, despite almost universal usage of supplemental oxygen therapy, the effects of different oxygenation levels under normobaric conditions on outcomes of patients presenting in the emergency department with TBI are unknown.

On the one hand, liberal oxygenation may provide a margin of safety against hypoxemia and may be needed to meet the high oxygen demands of an acutely altered brain physiology. On the other hand, there are increasing concerns that excessive oxygen supplementation may have harmful effects, such as central nervous system toxicity, cerebral vasoconstriction, impaired immunity leading to predisposition to infections (including pneumonia) and acute lung injury/acute respiratory distress syndrome. Such effects could be avoided by intermediate normal oxygen levels.

Taken together, the relative merits and risks of the abovementioned two approaches to oxygen therapy (namely, intermediate normal versus high normal oxygen levels) of patients with TBI in terms of important clinical outcomes (namely, development of nosocomial pneumonia, acute respiratory distress syndrome, disability and mortality) remain undefined. This suggests the need for randomized controlled trials. However, randomized controlled trials focusing on patient-centered outcomes should be preceded by pilot randomized controlled trials, which demonstrate a separation in treatment and protocol compliance (feasibility) associated with the studied interventions.

Therefore, the investigators propose a pilot multi-center randomized controlled trial to test the hypothesis that maintaining intermediate normal as opposed to high normal oxygen levels in patients presenting in the emergency department with TBI is feasible, and to obtain preliminary data on the efficacy of the two approaches to oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥18 years
* Glasgow Coma Scale ≤ 8
* Non-penetrating traumatic brain injury
* Intubated patient

Exclusion Criteria:

* Age <18 years
* Lack of intention to admit to the intensive care unit
* Moribund patient expected to die within 24 hours
* Expected need for mechanical ventilation < 24 hours
* Time interval from intubation to group allocation more than 60 minutes
* Penetrating traumatic brain injury
* Pregnancy
* Lack of equipoise of the treating clinician
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Mean area-under-curve (AUC) for SpO2 | Measurements will be obtained each hour for a total duration of 6 hours from intubation.
  SpO2 will be recorded each hour for a total duration of 6 hours from intubation. Subsequently, mean area-under-curve (AUC) will be calculated for each group. This will demonstrate the feasibility of the study.
Mean area-under-curve (AUC) for FiO2 | Measurements will be obtained each hour for a total duration of 6 hours from intubation.
  FiO2 will be recorded each hour for a total duration of 6 hours from intubation. Subsequently, mean area-under-curve (AUC) will be calculated for each group. This will demonstrate the feasibility of the study.
PaO2 | Measurements will be obtained at least once during 6 hours from intubation.
  PaO2 will be recorded at least once during 6 hours from intubation. Subsequently, PaO2 values (mmHg) will be calculated for each group. This will demonstrate the feasibility of the study.

SECONDARY OUTCOMES:
Nosocomial pneumonia | Within 7 days of subject enrollment
  Incidence of nosocomial pneumonia will be recorded for each arm
Acute Respiratory Distress Syndrome (ARDS) | Within 7 days of subject enrollment
  Incidence of ARDS will be recorded for each arm
All-cause mortality | Within 28 days of subject enrollment
  All-cause mortality will be recorded during ICU stay
Extended Glasgow Outcome Score (GOS-E) | At 6 months following subject enrollment
  A combined outcome of disability and mortality at 6 months using the Extended Glasgow Outcome Score will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ilias I Siempos, MD, DSc, Principal Investigator — Evangelismos Hospital, Athens, Greece
Locations (2):
- Greece (2):
  - Evangelismos Hospital, Athens
  - KAT General Hospital, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asehnoune K, Seguin P, Allary J, Feuillet F, Lasocki S, Cook F, Floch H, Chabanne R, Geeraerts T, Roger C, Perrigault PF, Hanouz JL, Lukaszewicz AC, Biais M, Boucheix P, Dahyot-Fizelier C, Capdevila X, Mahe PJ, Le Maguet P, Paugam-Burtz C, Gergaud S, Plaud B, Constantin JM, Malledant Y, Flet L, Sebille V, Roquilly A; Corti-TC Study Group. Hydrocortisone and fludrocortisone for prevention of hospital-acquired pneumonia in patients with severe traumatic brain injury (Corti-TC): a double-blind, multicentre phase 3, randomised placebo-controlled trial. Lancet Respir Med. 2014 Sep;2(9):706-16. doi: 10.1016/S2213-2600(14)70144-4. Epub 2014 Jul 24. PMID 25066331
- [Background] Asehnoune K, Balogh Z, Citerio G, Cap A, Billiar T, Stocchetti N, Cohen MJ, Pelosi P, Curry N, Gaarder C, Gruen R, Holcomb J, Hunt BJ, Juffermans NP, Maegele M, Midwinter M, Moore FA, O'Dwyer M, Pittet JF, Schochl H, Schreiber M, Spinella PC, Stanworth S, Winfield R, Brohi K. The research agenda for trauma critical care. Intensive Care Med. 2017 Sep;43(9):1340-1351. doi: 10.1007/s00134-017-4895-9. Epub 2017 Jul 29. PMID 28756471
- [Background] Dewan MC, Rattani A, Gupta S, Baticulon RE, Hung YC, Punchak M, Agrawal A, Adeleye AO, Shrime MG, Rubiano AM, Rosenfeld JV, Park KB. Estimating the global incidence of traumatic brain injury. J Neurosurg. 2018 Apr 27;130(4):1080-1097. doi: 10.3171/2017.10.JNS17352. Print 2019 Apr 1. PMID 29701556
- [Background] Andrews PJ, Sinclair HL, Rodriguez A, Harris BA, Battison CG, Rhodes JK, Murray GD; Eurotherm3235 Trial Collaborators. Hypothermia for Intracranial Hypertension after Traumatic Brain Injury. N Engl J Med. 2015 Dec 17;373(25):2403-12. doi: 10.1056/NEJMoa1507581. Epub 2015 Oct 7. PMID 26444221
- [Background] The Lancet Neurology. A rally for traumatic brain injury research. Lancet Neurol. 2013 Dec;12(12):1127. doi: 10.1016/S1474-4422(13)70266-7. No abstract available. PMID 24229612
- [Background] Xu F, Liu P, Pascual JM, Xiao G, Lu H. Effect of hypoxia and hyperoxia on cerebral blood flow, blood oxygenation, and oxidative metabolism. J Cereb Blood Flow Metab. 2012 Oct;32(10):1909-18. doi: 10.1038/jcbfm.2012.93. Epub 2012 Jun 27. PMID 22739621
- [Background] Vilalta A, Sahuquillo J, Merino MA, Poca MA, Garnacho A, Martinez-Valverde T, Dronavalli M. Normobaric hyperoxia in traumatic brain injury: does brain metabolic state influence the response to hyperoxic challenge? J Neurotrauma. 2011 Jul;28(7):1139-48. doi: 10.1089/neu.2010.1720. Epub 2011 Jun 30. PMID 21534719
- [Background] Tolias CM, Reinert M, Seiler R, Gilman C, Scharf A, Bullock MR. Normobaric hyperoxia--induced improvement in cerebral metabolism and reduction in intracranial pressure in patients with severe head injury: a prospective historical cohort-matched study. J Neurosurg. 2004 Sep;101(3):435-44. doi: 10.3171/jns.2004.101.3.0435. PMID 15352601
- [Background] Hafner S, Beloncle F, Koch A, Radermacher P, Asfar P. Hyperoxia in intensive care, emergency, and peri-operative medicine: Dr. Jekyll or Mr. Hyde? A 2015 update. Ann Intensive Care. 2015 Dec;5(1):42. doi: 10.1186/s13613-015-0084-6. Epub 2015 Nov 19. PMID 26585328
- [Background] Vincent JL, Taccone FS, He X. Harmful Effects of Hyperoxia in Postcardiac Arrest, Sepsis, Traumatic Brain Injury, or Stroke: The Importance of Individualized Oxygen Therapy in Critically Ill Patients. Can Respir J. 2017;2017:2834956. doi: 10.1155/2017/2834956. Epub 2017 Jan 26. PMID 28246487
- [Background] Raj R, Bendel S, Reinikainen M, Kivisaari R, Siironen J, Lang M, Skrifvars M. Hyperoxemia and long-term outcome after traumatic brain injury. Crit Care. 2013 Aug 19;17(4):R177. doi: 10.1186/cc12856. PMID 23958227
- [Background] Brenner M, Stein D, Hu P, Kufera J, Wooford M, Scalea T. Association between early hyperoxia and worse outcomes after traumatic brain injury. Arch Surg. 2012 Nov;147(11):1042-6. doi: 10.1001/archsurg.2012.1560. PMID 22801994
- [Background] Chu DK, Kim LH, Young PJ, Zamiri N, Almenawer SA, Jaeschke R, Szczeklik W, Schunemann HJ, Neary JD, Alhazzani W. Mortality and morbidity in acutely ill adults treated with liberal versus conservative oxygen therapy (IOTA): a systematic review and meta-analysis. Lancet. 2018 Apr 28;391(10131):1693-1705. doi: 10.1016/S0140-6736(18)30479-3. Epub 2018 Apr 26. PMID 29726345
- [Background] Panwar R, Hardie M, Bellomo R, Barrot L, Eastwood GM, Young PJ, Capellier G, Harrigan PW, Bailey M; CLOSE Study Investigators; ANZICS Clinical Trials Group. Conservative versus Liberal Oxygenation Targets for Mechanically Ventilated Patients. A Pilot Multicenter Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Jan 1;193(1):43-51. doi: 10.1164/rccm.201505-1019OC. PMID 26334785
- [Background] Robba C, Poole D, McNett M, Asehnoune K, Bosel J, Bruder N, Chieregato A, Cinotti R, Duranteau J, Einav S, Ercole A, Ferguson N, Guerin C, Siempos II, Kurtz P, Juffermans NP, Mancebo J, Mascia L, McCredie V, Nin N, Oddo M, Pelosi P, Rabinstein AA, Neto AS, Seder DB, Skrifvars MB, Suarez JI, Taccone FS, van der Jagt M, Citerio G, Stevens RD. Mechanical ventilation in patients with acute brain injury: recommendations of the European Society of Intensive Care Medicine consensus. Intensive Care Med. 2020 Dec;46(12):2397-2410. doi: 10.1007/s00134-020-06283-0. Epub 2020 Nov 11. PMID 33175276
- [Background] Busl KM. Nosocomial Infections in the Neurointensive Care Unit. Neurosurg Clin N Am. 2018 Apr;29(2):299-314. doi: 10.1016/j.nec.2017.11.008. PMID 29502719
- [Background] Girardis M, Busani S, Damiani E, Donati A, Rinaldi L, Marudi A, Morelli A, Antonelli M, Singer M. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1583-1589. doi: 10.1001/jama.2016.11993. PMID 27706466
- [Background] Siemieniuk RAC, Chu DK, Kim LH, Guell-Rous MR, Alhazzani W, Soccal PM, Karanicolas PJ, Farhoumand PD, Siemieniuk JLK, Satia I, Irusen EM, Refaat MM, Mikita JS, Smith M, Cohen DN, Vandvik PO, Agoritsas T, Lytvyn L, Guyatt GH. Oxygen therapy for acutely ill medical patients: a clinical practice guideline. BMJ. 2018 Oct 24;363:k4169. doi: 10.1136/bmj.k4169. No abstract available. PMID 30355567
- [Background] Mackle DM, Bailey MJ, Beasley RW, Bellomo R, Bennett VL, Deane AM, Eastwood GM, Finfer S, Freebairn RC, Litton E, Linke NJ, McArthur CJ, McGuinness SP, Panwar R, Young PJ; Australian and New Zealand Intensive Care Society Clinical Trials Group. Protocol summary and statistical analysis plan for the intensive care unit randomised trial comparing two approaches to oxygen therapy (ICU-ROX). Crit Care Resusc. 2018 Mar;20(1):22-32. PMID 29458318